CLINICAL TRIAL: NCT03873337
Title: Persistence Targeted Smoking Cessation in Schizophrenia (PTSC-S)
Brief Title: Persistence Targeted Smoking Cessation in Serious Mental Illness (SMI)
Acronym: PTSC-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marc L. Steinberg, Ph.D., Professor of Psychiatry, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018001696; R33DA041163 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2022-08-16 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-08

CONDITIONS: Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Tobacco Use Disorder; Schizophrenia; Schizoaffective Disorder
Keywords: tobacco; cigarette; schizophrenia; schizoaffective disorders; smoking cessation
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Tobacco Use Disorder; Schizophrenia; Psychotic Disorders; Smoking Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Due to the pandemic, this study was modified from a randomized clinical trial to test the feasibility, initial efficacy, and mechanisms of action of our PTSC-S intervention to a feasibility and acceptability test of our intervention when delivered via telehealth in a single group, within-subjects design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NRT + Persistence Targeted Smoking Cessation in SMI (Experimental): Participants will receive 10 weeks of nicotine patch (NRT) plus 8 weeks of task persistence focused cessation counseling delivered via telehealth.
  Interventions: Behavioral: Persistence Targeted Smoking Cessation in SMI (PTSC-S); Drug: Nicotine patch

INTERVENTIONS:
Behavioral: Persistence Targeted Smoking Cessation in SMI (PTSC-S) — All participants will receive 8 weeks of persistence focused smoking cessation counseling delivered via telehealth
Drug: Nicotine patch — All participants will receive 10 weeks of nicotine patch

SUMMARY:
Due to the pandemic, this study was modified from a randomized clinical trial to test the feasibility, initial efficacy, and mechanisms of action of our PTSC-S intervention to a feasibility and acceptability test of our intervention when delivered via telehealth in a single group, within-subjects design.

DETAILED DESCRIPTION:
The investigators will test the feasibility and acceptability of a telehealth-delivered treatment designed to help smokers with serious mental illness to quit using a therapy approach focused on increasing task persistence.

We will provide free, weekly individual telehealth video counseling sessions for 8 weeks and 10-weeks' worth of the nicotine transdermal patch (an FDA-approved smoking cessation product available over the counter). All sessions will be video recorded for treatment integrity and supervision.

The investigators hypothesize that 1) the PTSC-S intervention will be acceptable to participants, and the study will be feasible to conduct. We will report prolonged and point prevalence abstinence rates at end-of-counseling and at 3-month follow-up (CO verified <8ppm).

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18 - 70 years old
* Must indicate willingness to make a quit attempt in the next 30 days
* Must report being a daily cigarette smoker (including those labeled "little cigars") for past month
* Must have a diagnosis of Schizophrenia, Schizoaffective Disorder, or Bipolar Disorder on the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM), 5th edition, Research Version (SCID-5-RV)
* Psychiatric illness must be stable, as indicated by no hospitalizations in previous 8 weeks, and a stable psychotropic medication regimen for 8 weeks
* Must have a smartphone, tablet, or computer with ability to download apps
* Must currently receive mental health treatment
* Must sign release of information for current mental health treatment providers

Exclusion Criteria:

* Must not currently (in past 10 days) be taking varenicline (Chantix),
* Must not currently (in past 10 days) be taking bupropion (Zyban/Wellbutrin) to quit smoking.
* Must not be taking any nicotine preparations (gum, lozenge, patch, spray, inhaler) daily over the last 10 days
* Must not report myocardial infarction, unstable angina pectoris, or significant cardiac arrhythmia (including atrial fibrillation) in the past 30 days.
* Women must not be pregnant, "test positive" on a pregnancy test, nursing, or planning on becoming pregnant in the next three months. Women who can become pregnant may be included if using effective birth control.
* Must not have pending legal matters with potential to result in jail time
* Must not be planning on moving outside local area in next 3-months
* Problematic substance use in the past 3 months (Alcohol Use Disorders Identification Test-Concise (AUDIT-C) ≥5 for men and ≥4 for women, Drug Abuse Screening Test (DAST-10) score of ≥4)
* Must not have suicidal ideation in the past week with intent, plan, or access to method; must not have attempted suicide in the past year (as assessed on the SCID-RV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc L Steinberg, Ph.D., Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Division of Addiction Psychiatry, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for de-identified data from qualified researchers will be considered once the study has been completed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available once the study has been completed and primary and secondary outcomes have been published.
Access Criteria: Requests will be evaluated by the principal investigator. Access will be granted to the scientific researchers providing a valid scientific rationale for the request.

RESULTS

PARTICIPANT FLOW:
Groups:
- NRT + Persistence Targeted Smoking Cessation in Serious Mental Illness (SMI): Participants will receive 10 weeks of nicotine patch (NRT) plus 8 weeks of task persistence focused cessation counseling delivered via telehealth.
  Persistence Targeted Smoking Cessation in SMI (PTSC-S): All participants will receive 8 weeks of persistence focused smoking cessation counseling delivered via telehealth
  Nicotine patch: All participants will receive 10 weeks of nicotine patch
Period: Overall Study
Arm/Group | NRT + Persistence Targeted Smoking Cessation in Serious Mental Illness (SMI)
Started | 34
Completed | 22
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, Continuous (in years) as self reported by participants.
  years | 42.65 (11.96)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender Identity as self-reported by participants
  Participants
    Male | 16
    Female | 17
    Gender Nonconforming | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 22
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 34
relight [Count of Participants; unit: Participants] — Do you sometimes "butt out" or extinguish and re-light your cigarettes? (Yes/No)
  Participants
    Yes | 24
    No | 10

OUTCOME MEASURES:

1. Primary Outcome: Acceptability 1: Participant Rating of Usefulness of Intervention
Description: After each session, participants (N=33) provided a 1-7 rating of how "easy to understand" and how "helpful" the intervention was. Higher numbers represent greater ease and greater helpfulness, respectfully. There is no official scale title because the scale was developed for this study.
Time Frame: 3-months post quit date (approximately 4-months after baseline assessment)
Population: Participants who attended at least 1 counseling session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 33
units on a scale
  "Easy to understand" | 6.62 (0.95)
  "Helpful" | 6.58 (0.97)

2. Primary Outcome: Acceptability 2: Participant Rating of Counseling Session Length
Description: After each session, participants (N=33) provided a 1-7 rating of agreement with the statement, "There was too much information in today's session." (as a proxy for appropriateness of session length). Higher numbers represent greater agreement. There is no official scale title because the scale was developed for this study.
Time Frame: 3-months post quit date (approximately 4 months after baseline assessment)
Population: Participants who attended at least one counseling session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 33
units on a scale | 2.29 (1.93)

3. Primary Outcome: Acceptability 3: Participant Rating of Treatment Length / Timing of Target Quit-Date
Description: We asked participants how acceptable the placement of the target quit date was to participants (i.e., it was scheduled for session 4). We report the percentage of participants who responded that the quit date was "too soon", "too late", or "just about right".
Time Frame: 3-months post quit date (approximately 4 months after baseline assessment)
Population: Participants who responded to the item regarding acceptability of setting the target quit date for the 4th session.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 28
Participants
  4th session was too soon | 14
  Fourth session was too late | 2
  Fourth session was at just about the right time. | 12

4. Primary Outcome: Feasibility 1: Number of Participants Contacted at 3 Months Post-Quite Date
Description: We will calculate follow-up rates to determine if they meet our goal of 80% follow-up rates at the 3-month follow-up.
Time Frame: 3-months post quit date (approximately 4 months after baseline assessment)
Population: Participants enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Participants | 28

5. Primary Outcome: Feasibility 2: Missing/Unusable Data
Description: We will determine the rate of missing or unusable carbon monoxide (CO) data to determine if the rate meets our goal of less than 10% missing/unusable data. There were a possible 340 CO assessment data points.
Time Frame: 3-months post quit date (approximately 4 months after baseline assessment)
Population: 340 potential CO data points (Participants enrolled in the study (N=34) with a potential 10 CO assessments each = 340 potential CO data points)
Measure: Number; unit: Missing CO points (out of 340)
Units Other Than Participants: CO assessment data points
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Number analyzed (CO assessment data points) | 340
Missing CO points (out of 340) | 184

6. Primary Outcome: Feasibility 3: Participant Attendance
Description: Participants in the PTSC-S intervention will attend at least 60% of their sessions
Time Frame: 8 weeks of counseling with a 2-week grace period to make up missed sessions (10 weeks)
Population: All participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Participants
  Attended 0 of 8 counseling sessions | 1
  Attended 1 of 8 counseling session | 2
  Attended 2 of 8 counseling sessions | 5
  Attended 3 of 8 counseling sessions | 4
  Attended all 8 counseling sessions | 22

7. Secondary Outcome: Number of Participants With Seven-day Point Prevalence Abstinence at End-of-counseling
Description: No smoking on the 7 days before the final counseling session, biochemically verified with CO<8ppm
Time Frame: End-of-counseling (8 weeks)
Population: Participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Participants | 3

8. Secondary Outcome: Number of Participants With Prolonged Abstinence at End-of-counseling
Description: Prolonged abstinence with a 2-week grace period following the target quit date until end-of-counseling, biochemically verified with CO<8ppm
Time Frame: End-of-counseling (8 weeks)
Population: Participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Participants | 2

9. Secondary Outcome: Number of Participants With Seven-day Point Prevalence Abstinence at 3-month Follow-up
Description: No smoking on the 7 days before the 3-month follow-up, biochemically verified with CO<8ppm
Time Frame: 3-months post target quit date (approximately 4 months after baseline assessment)
Population: Participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Participants | 3

10. Secondary Outcome: Number of Participants With Prolonged Abstinence at at 3-month Followup
Description: Prolonged abstinence with a 2-week grace period following the target quit date until 3-months post quit-date, biochemically verified with CO<8ppm
Time Frame: 3-months post target quit date (approximately 4 months after baseline assessment)
Population: Participants enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 34
Participants | 2

11. Secondary Outcome: Task Persistence Scores
Description: 14-item Thoughts About Smoking Questionnaire (TASQ). Lower scores represent greater task persistence. The total score can range from a minimum of 14 to a maximum of 98.
Time Frame: 2 months after baseline assessment and 4 months after baseline assessment
Population: Participants for whom we have baseline and 2-months post-baseline data (n=26) and 4-months post-baseline data (n=28).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 28
units on a scale
  2 months post-baseline: number analyzed (Participants) | 26
  2 months post-baseline | 44.19 (21.72)
  4 months post-baseline | 47.39 (26.34)
Statistical Analysis 1: Comparison: NRT + Persistence Targeted Smoking Cessation in SMI; One-tailed, paired sample t-tests will be used to examine decreases in scores on the TASQ at one-month post target quit date (2-months after baseline assessment; Test type: Superiority; p < 0.001, t-test, 1 sided — not adjusted for multiple comparisons; df = 25
Statistical Analysis 2: Comparison: NRT + Persistence Targeted Smoking Cessation in SMI; One-tailed, paired sample t-tests will be used to examine decreases in scores on the TASQ at 3-months post target quit date (4 months after baseline assessment; Test type: Superiority; p = 0.002, t-test, 1 sided — not adjusted for multiple comparisons; df = 27

12. Secondary Outcome: Cigarettes Per Day
Description: Hypothesis 3: As compared to baseline, participants will report smoking fewer cigarettes per day at 2- and 4-months post-baseline. Analysis 3: One-tailed, paired sample t-tests will be used to examine decreases in cigarettes smoked per day on the TASQ at each timepoint.
Time Frame: 2 months after baseline assessment and 4 months after baseline assessment
Population: Number of participants for whom we had data for mean cigarettes per day in the preceding week at baseline and 2 months post-baseline and at baseline and 4-months post-baseline.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
Number analyzed (Participants) | 28
cigarettes per day
  2 months post-baseline | 7.01 (8.34)
  4 months post-baseline | 8.48 (9.31)
Statistical Analysis 1: Comparison: NRT + Persistence Targeted Smoking Cessation in SMI; One-tailed, paired sample t-tests will be used to examine decreases in cigarettes smoked per day at one-month post target quit date (2-months after baseline assessment; Test type: Superiority; p < 0.001, t-test, 1 sided — not adjusted for multiple comparisons; df = 27
Statistical Analysis 2: Comparison: NRT + Persistence Targeted Smoking Cessation in SMI; One-tailed, paired sample t-tests will be used to examine decreases in cigarettes smoked per day at 3-months post target quit date (4-months after baseline assessment; Test type: Superiority; p < 0.001, t-test, 1 sided — not adjusted for multiple comparisons; df = 27

ADVERSE EVENTS:
Time Frame: Four months
Arm/Group | NRT + Persistence Targeted Smoking Cessation in SMI
All-Cause Mortality (participants affected / at risk) | 2/34
Serious Adverse Events (participants affected / at risk) | 3/34
Other Adverse Events (participants affected / at risk) | 19/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRT + Persistence Targeted Smoking Cessation in SMI (N=34)
Fractured nose (Injury, poisoning and procedural complications) | 1 (1) — Fall resulting in a fractured nose
Psychiatric hospitalization (Psychiatric disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NRT + Persistence Targeted Smoking Cessation in SMI (N=34)
skin irritation at the patch site (Skin and subcutaneous tissue disorders) | 4 (4)
Nausea / Upset stomach (Gastrointestinal disorders) | 3 (3)
Depression (Psychiatric disorders) | 10 (11)
Anxiety (Psychiatric disorders) | 6 (6)
Cold symptoms (Infections and infestations) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
Vivid dreams (Nervous system disorders) | 2 (2)
Increased psychiatric symptoms (Psychiatric disorders) | 6 (6) — Increased psychotic symptoms and/or increased agitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT03873337/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/37/NCT03873337/ICF_000.pdf